CLINICAL TRIAL: NCT01048138
Title: Use of Biperiden as a Disease Modifying Agent After Traumatic Brain Injury: a Placebo Controlled, Randomized, Double Blind Study
Brief Title: Use of Biperiden for the Prevention of Post-traumatic Epilepsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment and funding issues, together with the event of the SARS-CoV-2 pandemic prompted an adjustment in the study design to stop enrollment at 123 patients.
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luiz Eugenio Mello, Full Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP0560/05
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Traumatic Brain Injury
Keywords: Biperiden; Post-traumatic Epilepsy; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Epilepsy, Post-Traumatic | interventions — biperiden lactate; Biperiden; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biperiden Lactate (Experimental): 5mg IV(in the vein)every 6 hours for 10 days
  Interventions: Drug: Biperiden Lactate
- Placebo (Placebo Comparator): 5mg IV(in the vein)every 6 hours for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Biperiden Lactate — 5mg IV(in the vein)every 6 hours for 10 days
  Other Names: akineton; cinetol
  Arms: Biperiden Lactate
Drug: Placebo — 5mg IV(in the vein)every 6 hours for 10 days
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
There is no AED or medication that has been demonstrated to affect the development of post-traumatic epilepsy. Biperiden is a cholinergic antagonist, acting in the muscarinic receptor, that is widely used as an anti Parkinson drug. The investigators data with animal models of epilepsy indicate that anti-muscarinic agents might affect the natural course of the disease in the case of post-traumatic epilepsy.

DETAILED DESCRIPTION:
Treatment with biperiden should be initiated in the first 12 hours after trauma as means to avoid the epileptogenic process. The treatment will be repeated every 6 hours for 10 consecutive days. The efficacy of biperiden as an antiepileptogenic drug will be established by analyzing the development of PTE between the biperiden and placebo groups. Several patients' aspects (clinical, electroencephalography, brain imaging, genetic and behavioral data) will be monitored for two year follow-up to unravel the mechanisms by which biperiden exerts its actions on epileptogenesis. The investigators are already at the early stages of patient's recruitment using the available resources.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 75 year of age
* patients with a diagnosis of acute TBI admitted to an emergency unit within 12 hours of the accident, regardless of the accident
* brain CT scan with signs of acute intraparenchymatous contusion
* signed informed consent (possibly by a relative)

Exclusion Criteria:

* malignant neoplasia and other severe comorbidities
* neurodegenerative disorders
* previous cerebrovascular accident
* record of convulsive seizures or use of anti-epileptic medication
* pregnancy
* concomitant use of the other anticholinergic medications
* presence of any factor that may contraindicate the use of biperiden
* participation in other clinical trial
* alcohol intoxication will not lead to exclusion of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome: Indidence of post-traumatic epilepsy | 24 months after TBI
  The incidence of seizures will be evaluated starting immediately after TBI and continuously during the hospitalization period and after hospital discharge during the two year follow up period. Patients and their relatives will be asked to maintain a diary of seizures, and thus record all seizures with detailed descriptions of each event. The recordings will be evaluated in each patient visit. Seizures incidence will be compared between placebo and biperiden-treated patients.

SECONDARY OUTCOMES:
Frequency of seizures | 24 months after TBI
  The frequency of seizures will be counted starting immediately after TBI and continuously during the hospitalization period and after hospital discharge during the two year follow up period. Frequency of seizure will be compared between placebo and biperiden-treated patients.
Mortality and adverse effects | 24 months after TBI
  The incidence of death and adverse effects will be counted starting immediately after TBI and continuously during the hospitalization period and after hospital discharge during the two year follow up period. Incidence of death and adverse effects will be compared between placebo and biperiden-treated patients.

OTHER OUTCOMES:
Electroencephalogram Analysis: Presence of Epileptiform Discharges | during first 10 days after TBI and 1, 3, 6, 9, 12, 18 and 24 months after TBI
  Given the requirement of specific adjustments in the EEG recording apparatus (10 KHz sampling rate, high-pass filter above 80 Hz for ripples and 250 Hz for fast ripples), only a subset of patients will be included in this outcome. EEG will be continuously registered during the first 10 days after TBI, weekly until hospital discharge and at specified time frames after TBI. The presence of high frequency oscillations (ripples and fast ripples) will be investigated.
Cognitive Assessments - Wechsler Adult Intelligence Scale (WAIS) - III | 6, 12 and 24 months after hospital discharge
  Cognitive effects of the biperiden therapy will be assessed to demonstrate the efficacy and safety of this medicine in face of its possible cognitive implications. The instruments selected to assess those are tests of the Wechsler Adult Intelligence Scale (WAIS) - III. The WAIS-III returns scores on four separate indexes of adult intelligence, the Perceptual Reasoning Index, the Verbal Comprehension Index, the Working Memory Index and the Processing Speed Index. Scores will be calculated on each of the 4 indices and then combined to create a Full-Scale IQ. The WAIS-III is normed so that 100 is the median score for the adult population (score ranges: 120-129= superior, 110-119= high average, 90-109=average, 80-89= low average, 71-80= borderline intellectual functioning, 50-70= moderate retardation, below 50= severe retardation. The battery of tests will be applied at specific time frames and results will be compared.
Quality of Life assessments - European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L), EQ-VAS | 24 month after TBI
  The Brazilian version of the EQ-5D-3L and EQ-VAS questioner will be used to assess health-related quality of life (HRQoL), 24 months after TBI. It consists of a questionnaire covering five dimensions of HRQoL (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual analog scale (VAS). The descriptive system defines 243 different health states.
Blood sampling biomarkers - Expression of miRNAs | 10 days or 18 months after TBI
  Alterations in expression of miRNAs will be assayed in blood samples during treatment with biperiden, or 18 months after trauma. Patterns of changes in the miRNA levels will be compared between the groups of patients that developed post-traumatic epilepsy or did not develop epilepsy.
Blood sampling biomarkers - Expression of the ApoEϵ4 allele | 10 days or 18 months after TBI
  To investigate the expression of the ApoEϵ4 allele in TBI patients, and its correlation with post-traumatic epilepsy development and the biperiden treatment efficacy to prevent epilepsy, RFLP-PCR will be assayed in blood samples of TBI patients. The genotyping reactions will be performed blinded to clinical features. The presence of the ApoEϵ4 allele will be correlated with the incidence of seizures in the follow up assessments after TBI.
Blood sampling biomarkers - Expression of inflammatory cytokines | 10 days after TBI
  To verify whether cytokines are differently involved on PTE development, we will perform multi-analyte protein profile in blood plasma samples collected during treatment with biperiden. Simultaneous measuring of different proteins in plasma will be performed. The concentration of each analyte will be normalized to the total protein concentration and presented as a proportion of specific proteins in picograms (pg) per microgram (μg) of total protein. Patterns of protein expression will be correlated with the incidence of seizures in the follow up assessments after TBI.
Brain Activity Biomarkers - Presence of high frequency oscillations | during first 10 days after TBI and 1, 3, 6, 12, 18 and 24 months after TBI
  Given the requirement of specific adjustments in the EEG recording apparatus (10 KHz sampling rate, high-pass filter above 80 Hz for ripples and 250 Hz for fast ripples), only a subset of patients will be included in this outcome. EEG will be continuously registered during the first 10 days after TBI, weekly until hospital discharge and at specified time frames after TBI. The presence of high frequency oscillations (ripples and fast ripples) will be investigated.
Brain Activity Biomarkers - Presence of cortical spreading depression | during first 10 days after TBI
  Given the requirement of specific adjustments in the EEG recording apparatus (e.g., direct current [DC] recording) to detect cortical spreading depression, a subset of patients will be EEG continuously registered during the first 10 days after trauma with other recording specifications. The presence of cortical spreading depression activity will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Mello, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Foresti ML, Garzon E, de Moraes MT, Valeriano RPS, Santiago JP, Dos Santos GM, Longo NM, Baise C, Andrade JCQF, Susemihl MA, Leite CDC, Naffah Mazzacoratti MDG, Paiva WS, de Andrade AF, Teixeira MJ, Mello LE. Initial clinical evidence on biperiden as antiepileptogenic after traumatic brain injury-a randomized clinical trial. Front Neurol. 2024 Aug 7;15:1443982. doi: 10.3389/fneur.2024.1443982. eCollection 2024. PMID 39175759